CLINICAL TRIAL: NCT06384092
Title: Standardization of UV Exposure Methods (Artificial Source vs. Sunlight) in Dermatological Research: A Comprehensive Investigation Into the Efficacy Assessment Methodology for Anti-tanning Agents Through Process Validation
Brief Title: Process Validation in Dermatology: Assessing Methods for UV Exposure (Artificial Source vs. Sunlight) and Efficacy Evaluation of Anti-Tanning Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Principal Investigator, Maheshvari Patel, Principal Investigator - Director (Operations), NovoBliss Research Pvt Ltd
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NB240005-NB-V
Record Dates: First submitted 2024-02-06; First posted 2024-04-25 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Skin Pigmentation
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: Proof of science/concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Site T1 (Experimental): Test Product A - Test Sun Protection Cream Dosage Form - Cream Route of Administration - Topical Mode of Usage - Apply directly on the designated site till absorbed. Dosage - 0.2 mL/site
  Interventions: Other: Test Sun Protection Cream
- Site T2 (Active Comparator): Test Product B - Benchmark (Sun Protection Cream) Dosage Form - Cream Route of Administration - Topical Mode of Usage - Apply directly on the designated site till absorbed. Dosage - 0.2 mL/site
  Interventions: Other: Benchmark Sun Protection Cream
- Site U1-4 (No Intervention): Test Product : No test product applied.

INTERVENTIONS:
Other: Test Sun Protection Cream — Apply directly on the designated site till absorbed.
  Other Names: Test Treatment A
  Arms: Site T1
Other: Benchmark Sun Protection Cream — Apply directly on the designated site till absorbed.
  Other Names: Test Treatment B
  Arms: Site T2

SUMMARY:
The rationale of this study is to establish a robust method for assessing sun protection product efficacy in preventing erythema and tanning. Employing both artificial ultraviolet-A Irradiation and natural direct sunlight exposure, the investigation seeks to provide a reliable methodology, ensuring reproducibility and enabling a direct comparison between these methods. Meticulously determining optimal UV dosages, the study prioritizes inducing skin responses for evaluation while avoiding adverse effects like blistering. The localized validation of UV exposure techniques, tailored to the Indian population, contributes significantly to the field by addressing diverse skin types and environmental conditions. By incorporating both artificial and natural (direct sunlight) UV exposure methods, the study aspires to enhance the safety and effectiveness of future dermatological investigations, benefiting both the scientific community and the broader population.

ELIGIBILITY:
Inclusion Criteria:

1. 06 Healthy adult subjects aged between 18 to 45 years (both inclusive).
2. Healthy adult male and non-pregnant|non-lactating females.
3. Female of childbearing potential have self-reported negative urine pregnancy test.
4. Subjects with Fitzpatrick skin types III to V will be included. Alternatively, subjects with a Skin colorimetric Individual Typology Angle (ITA) value ranging from 20° to 41° at the application site (forearms) to be included to ensure a diverse representation of skin tones.
5. Absence of known photosensitivity disorders to maintain the integrity of the study outcomes.
6. Subjects must exhibit a willingness to comply with study plan, including follow-up visits and product applications.
7. No history of skin cancer to or any adverse skin conditions, and not under any medication(s) likely to interfere with the study results.
8. Subjects willing to follow study direction and willing to give written informed consent for the participation.

Exclusion Criteria:

1. Active skin diseases, such as eczema or psoriasis, that could potentially influence skin reactions.
2. Use of photosensitizing medications that interfere with UV-induced skin responses.
3. Pregnancy or breastfeeding status, as hormonal changes during these periods can affect skin reactions.
4. Individuals with a history of severe adverse reactions to skincare or cosmetic products, ensuring participant safety.
5. Presence of open wounds, infections, or cuts at the application sites to prevent complications during the study.
6. Subjects with a history of significant sunburns in the past three months, minimizing the potential for confounding effects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in Melanine index using instrumental assessment | Days 1, 3 and 7.
  Change in melanin index (MI) before and after the exposure as measured using the Changes in melanin index will be measured by using Mexameter® MX 18.
Change in erythema index using instrumental assessment | Days 1, 3 and 7.
  Change in the erythema index (EI) before and after the exposure as measured using the Mexameter® MX 18.

SECONDARY OUTCOMES:
Change in skin erythema/dryness/wrinkles and oedema using draize scale | Days 1, 3 and 7.
  Visual change in skin erythema/dryness/wrinkles and oedema of the skin using the Draize scale. Where 0=No reaction, 4=severe erythema/wrinkle/oedema

CONTACTS AND LOCATIONS:
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No